CLINICAL TRIAL: NCT03468621
Title: Relation of Skin Closure Method to Groin Wound Infections After Proximal Femoral Artery Exposure, a Randomized Clinical Trial
Brief Title: Relation of Skin Closure Method to Groin Wound Infections After Proximal Femoral Artery Exposure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Veikko Nikulainen, Resident in Vascular Surgery, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: National Wound Infection Study
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Surgical Wound Infection
Keywords: woundclosure; technique; surgical; site; infection; intrademal; transdermal; suture
MeSH Terms: conditions — Surgical Wound Infection; Infections

STUDY DESIGN:
Intervention Model Description: Patients are randomised to intradermal and transdermal wound closure techniques. Randomisation is 1:1 and block randomisation is used
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradermal wound closure (Other): Intradermal wound closure of the groin wound
  Interventions: Procedure: Wound closure
- Transdermal wound closure (Other): Wound closure of the groin wound with metal staples
  Interventions: Procedure: Wound closure

INTERVENTIONS:
Procedure: Wound closure — Method of wound closure
  Other Names: Intradermal wound closure; Transdermal wound closure

SUMMARY:
This study aims to asses whether the rate of surgical wound infections in vascular surgery procedures involving exposure of the proximal femoral artery can be reduced using a different skin closure technique.

DETAILED DESCRIPTION:
Summary of the research plan

Background - According to published articles the frequency of groin wound infections after peripheral revascularization varies substantially depending on the source from 5% up to 27%.

Aims of the study - The aim of this randomized clinical trial is to evaluate whether the number of groin wound infections can be reduced with an intradermal skin suture compared to the commonly used metal staples skin closure method.

Methods and study design - This is a randomized clinical trial of patients undergoing a vascular procedure which includes an incision in the groin. The patients will be randomized (1:1) to two different wound closure techniques: subcuticular suture or metal staples. After the procedure the patients will be controlled for four to six weeks and the infection rate in each group is recorded. A clinical diagnosis of infection according to Centre for Disease Control (CDC) guidelines will be recorded, no microbiological samples will be routinely collected.

Statistical analysis - A power analysis has been conducted based on Finnish RCT studies and a retrospective study from our own hospital (submitted to Annals of Vascular Surgery 1/2018) which included all isolated groin wounds from Turku University Hospital Vascular Surgery clinic 2015-2016. According to this analysis between 130-150 patients are needed for each group.

Time and schedule- This is a multicenter trial. Ethical committee approval was acquired in 2015. The randomization will start in the spring of 2018 in the University Hospital of Turku. Later in the year in the other hospitals that are participating in the study once the regional authorities have given their consent.

Ethical aspects - Ethical committee approval was obtained in 2015. The wound closure techniques are all in everyday use already, nothing new and experimental will be used.

Budget - This study is a critical part of quality control and improvement in vascular surgery. The funding will be applied from the Finnish Academy and EVO funding from the ERVA.

ELIGIBILITY:
Inclusion Criteria:

* Primary procedure to the groin, isolated groin wound

Exclusion Criteria:

* Emergency procedure, secondary procedure, wound is a part of a larger wound in the same limb

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
SWI | 4-6weeks from surgery
  Surgical wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Harri Hakovirta, adj prof., Study Director — harri hakovirta@tyks.fi
Locations (3):
- Finland (3):
  - Keski-Suomen keskussairaala, Jyväskylä, Central Finland
  - Satakunnan keskussairaala, Pori, Satakunta
  - University Hospital of Turku, Turku, Southwest Finland

IPD SHARING:
Plan to Share IPD: No
Due to European and Finnish legislation. The information of individual patients is not possible By other researchers.

REFERENCES:
- [Background] Turtiainen J, Saimanen E, Partio T, Karkkainen J, Kiviniemi V, Makinen K, Hakala T. Surgical wound infections after vascular surgery: prospective multicenter observational study. Scand J Surg. 2010;99(3):167-72. doi: 10.1177/145749691009900312. PMID 21044935
- [Background] Derksen WJ, Verhoeven BA, van de Mortel RH, Moll FL, de Vries JP. Risk factors for surgical-site infection following common femoral artery endarterectomy. Vasc Endovascular Surg. 2009 Feb-Mar;43(1):69-75. doi: 10.1177/1538574408323502. Epub 2008 Sep 30. PMID 18829586
- [Background] Daryapeyma A, Ostlund O, Wahlgren CM. Healthcare-associated infections after lower extremity revascularization. Eur J Vasc Endovasc Surg. 2014 Jul;48(1):72-7. doi: 10.1016/j.ejvs.2014.02.003. Epub 2014 Mar 6. PMID 24613135
- [Background] Stewart AH, Eyers PS, Earnshaw JJ. Prevention of infection in peripheral arterial reconstruction: a systematic review and meta-analysis. J Vasc Surg. 2007 Jul;46(1):148-55. doi: 10.1016/j.jvs.2007.02.065. PMID 17606135
- [Background] Murphy PG, Tadros E, Cross S, Hehir D, Burke PE, Kent P, Sheehan SJ, Colgan MP, Moore DJ, Shanik GD. Skin closure and the incidence of groin wound infection: a prospective study. Ann Vasc Surg. 1995 Sep;9(5):480-2. doi: 10.1007/BF02143863. PMID 8541198
- [Background] Gurusamy KS, Toon CD, Allen VB, Davidson BR. Continuous versus interrupted skin sutures for non-obstetric surgery. Cochrane Database Syst Rev. 2014 Feb 14;2014(2):CD010365. doi: 10.1002/14651858.CD010365.pub2. PMID 24526375
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585
- [Derived] Nikulainen V, Helmio P, Salminen P, Hurme S, Kukkonen T, Koskinen T, Hakovirta H. Effect of Skin Closure with Metal Staples vs. Intradermal Suture on Groin Infections after Vascular Surgery: A Randomised Controlled Trial. Eur J Vasc Endovasc Surg. 2025 May;69(5):777-782. doi: 10.1016/j.ejvs.2025.02.004. Epub 2025 Feb 7. PMID 39923834

DOCUMENTS (1):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03468621/Prot_000.pdf